CLINICAL TRIAL: NCT01924741
Title: International Registry to Assess Outcomes of Major Liver Resections Requiring Two Interventions Including the New Operation Associating Liver Partition With Portal Vein Ligation for Staged Hepatectomy (ALPPS)
Brief Title: Registry of Major Liver Resections Including ALPPS and Other Liver Resections in Two Stages
Acronym: ALPPSREG
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: ALPPS registry
Record Dates: First submitted 2013-08-14; First posted 2013-08-16 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Liver Neoplasms; Liver Regeneration
Keywords: Liver neoplasms; Liver regeneration
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALPPS: ALPPS is the most recent modification of the techniques developed for Two-stage hepatectomies. ALPPS allows to remove an extensive part of the liver in two steps. In the first step the liver parenchyma is transected along the intended line of resection and the future liver remnant cleaned by partial resections from all tumor tissue in the case of bilobar tumors. To this a portal ligation of the larger liver lobe that will have to be removed is added. After a waiting period of 1-2 weeks the second step is performed in which the deportalized liver is removed to render the patient completely tumor-free. (Ann Surg 2012; 255(3):405-14.)
  Interventions: Procedure: ALPPS

INTERVENTIONS:
Procedure: ALPPS — Other procedures related to ALPPS like banding of the parechyma with portal vein ligation etc.
  Other Names: In-situ split hepatectomy

SUMMARY:
Recently a new method of induce similar hypertrophy in the liver as is observed after hepatectomy has been described and was given the eponym "ALLPS". "ALPPS" stands for Associating Liver Partition with Portal Vein Ligation for Staged Hepatectomy (ALPPS).

Since the procedure is used worldwide this international registry was created to enable tracking of cases performed worldwide for safety and outcomes and innovations by the groups involved as well as allows a non-randomized comparison to the conventional methods of portal vein occlusion.

DETAILED DESCRIPTION:
The ALPPS registry is accessible online through the data portal www.allps.net. Registered members recieve access through a member ID and password. Data submission is supported by the SECUTRIAL software, supported by the Clinical Trials center of the University of Zurich.

All data submitted are anonymized before entry through the SECUTRIAL Software. Administration of the registry data is performed through the Department of Visceral and Transplantation Surgery in the University Hospital Zurich and the Clinical Trials Center of the University of Zurich, Switzerland, in collaboration with the Italian Hospital in Buenoas Aires, Argentina.

A Scientific Committee has been appointed to give approval for any data analysis. Any participating center may apply for data analysis.

Particiating International Centers have responsibility for the validity of the data submitted and the respective local institutional review procedures.

ELIGIBILITY:
Inclusion Criteria:

* All Patients who undergo the new ALPPS procedure
* Patients undergoing any other modification of ALPPS like portal vein embolization (PVE) or banding of the liver with portal vein ligation or embolisation or other liver resection in two stages resembling ALPPS_
* Male and Female patients 18 years to no limit
* Prior registering the data, patient was informed and did not object to the use of his/her anonymized medical data in this registry

Exclusion Criteria:

* No exclusion criteria apply for a registry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primarily non-resectable liver tumors
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Morbidity and mortality (peripoerative) | 3 months
  Primary outcome variablesis perioperative mortality and complications and survival status after 3 months. Data will be entered following the widely accepted Clavien-Dindo classification system .

SECONDARY OUTCOMES:
Long term survival | 5 years
  Outcome variables include long term survival after 3, 6, 12, 18 and 24 month, survival status after 3, 4, and 5 years. If the patient is still alive the data about hepatic recurrence and systemic recurrence will be collected. If there is a recurrence the type of treatment will be recorded.
Perioperative liver and renal function | 5 days
  Outcome variables include liver and renal function after surgery. INR and Total bilirubin as well as creatinine prior to surgery and 5 days after stage 1 and five days after stage 2 are recorded and commonly accepted citeria for postoperative liver and postoperative renal failure are used to assess these 2 types of complications.
Disease specific recurrence/failure to cure | 5 years
  Outcome variables include disease specific failure to cure (to completely resect) or disease specific recurrence after 3, 6, 12, 18 and 24 month, survival status after 3, 4, and 5 years. If there is a failure to cure or recurrence, the type of treatment will be recorded.
Liver Growth as assessed by imaging-based volumetry | between stage 1 and stage 2 (1-12 weeks)
  Outcomes variables include Liver Growth as assessed by imaging-based volumetry between stage 1 and stage 2 (1-12 weeks)as assessed either by computer tomography or magnetic resonance based volumetry

OTHER OUTCOMES:
Inclusion criteria by registry participants | at enrollment
  The registry will evaluate the criteria used by study participants to include patients to the ALPPS procedure including tumor type, size, number extent, liver parechymal quality, starting volumes, resection volumes and specific methods of resection or sequneces of methods of resection used.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alain Clavien, Prof, MD, PhD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Background] Schnitzbauer AA, Lang SA, Goessmann H, Nadalin S, Baumgart J, Farkas SA, Fichtner-Feigl S, Lorf T, Goralcyk A, Horbelt R, Kroemer A, Loss M, Rummele P, Scherer MN, Padberg W, Konigsrainer A, Lang H, Obed A, Schlitt HJ. Right portal vein ligation combined with in situ splitting induces rapid left lateral liver lobe hypertrophy enabling 2-staged extended right hepatic resection in small-for-size settings. Ann Surg. 2012 Mar;255(3):405-14. doi: 10.1097/SLA.0b013e31824856f5. PMID 22330038
- [Derived] Reese T, Fard-Aghaie MH, Makridis G, Kantas A, Wagner KC, Malago M, Robles-Campos R, Hernandez-Alejandro R, de Santibanes E, Clavien PA, Petrowsky H, Linecker M, Oldhafer KJ. Renal Impairment Is Associated with Reduced Outcome After Associating Liver Partition and Portal Vein Ligation for Staged Hepatectomy. J Gastrointest Surg. 2020 Nov;24(11):2500-2507. doi: 10.1007/s11605-019-04419-2. Epub 2019 Nov 19. PMID 31745902
- See also: Click here to receive more information about ALPPS registry and studies — http://www.alpps.net